CLINICAL TRIAL: NCT03754803
Title: Description of Real World Antiviral Effectiveness and Sustainability of the 2-Drug Regimen Dolutegravir + Lamivudine in Untreated and Pre-treated Patients in Routine Clinical Care in Germany
Acronym: URBAN
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: MUC Research GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 208983
Record Dates: First submitted 2018-10-11; First posted 2018-11-27 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: Dolutegravir; Two-drug regimen; Human Immunodeficiency Virus; HIV Symptom Distress Module; Lamivudine; HIV treatment satisfaction questionnaire
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — SDM; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total participants: Antiretroviral treatment (ART) naïve and pre-treated HIV-1 positive participants for whom DTG+3TC is indicated according to local label.
  Interventions: Other: HIV symptom distress module (SDM) questionnaire; Other: HIV treatment satisfaction questionnaire (TSQ)

INTERVENTIONS:
Other: HIV symptom distress module (SDM) questionnaire — The SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment.
Other: HIV treatment satisfaction questionnaire (TSQ) — The HIV TSQ is a 10-item-self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience and flexibility.

SUMMARY:
This is a prospective, non-interventional, multi-center study, in participants with clinical indication of Human Immunodeficiency Virus (HIV)-1 infection. The aim of the study was to generate the real world evidence for the use of DTG+3TC in routine clinical care in Germany to supplement data obtained from controlled clinical trials. Treatment naïve and pre-treated HIV-1 positive participants were enrolled in the study. The observation period for the study was 3 years. Data was collected from routine clinical care via electronic data capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

* Participants >= 18 years of age.
* Participants with documented HIV-1 infection.
* Prescription of DTG + 3TC was issued independently from entering this study.
* Participants with the ability to understand informed consent form and other relevant regulatory documents.

Exclusion Criteria:

* Any contraindication according to Tivicay or Lamivudine summaries of product characteristics (SmPCs).
* Participants with VL > 500 c/mL.
* Any antiretroviral therapy for the treatment of HIV-1 in addition to DTG and 3TC or the DTG/3TC fixed dose combination (FDC).
* Participants with hepatitis B virus (HBV)- coinfection.
* Participants with current participation in the ongoing non-interventional study TRIUMPH (study number: 202033, NCT number: NCT02342769) or in any interventional clinical trial irrespective of indication.
* Participants who had previously participated in clinical trials assessing DTG+ 3TC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naïve and pre-treated HIV-1 positive participants from Germany were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (9):
- Germany (9):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bochum
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
  - GSK Investigational Site, Osnabrück
  - GSK Investigational Site, Weimar

IPD SHARING:
Plan to Share IPD: No
Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.ViiV-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Under EU privacy laws, participants who withdraw consent can choose whether their data up to withdrawal may be used or must be deleted. Safety data (e.g., ADRs, SAEs) are exempt and must be retained. This resulted in a higher number of participants analyzed for the Safety Analysis Set (N = 368) compared to Effectiveness Analysis Set (N = 366).
Pre-assignment Details: A total of 376 participants were enrolled in the Full Analysis Set, of which 10 were excluded for various reasons, including protocol violations and participant withdrawal. The remaining 366 participants were included in the Effectiveness Analysis Set.
Period: Overall Study
Arm/Group | Total Participants
Started (Safety Analysis Set) | 368
Effectiveness Analysis Set | 366
Completed | 366
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The Baseline analysis was performed on the Effectiveness Set which includes all participants from the Full Analysis Set except those excluded for various reasons, such as protocol violations and participant withdrawal.
Arm/Group | Total Participants
Number analyzed (Participants) | 366
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 47.0 [38.0 to 54.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 341
  Female | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Low Level Viremia
Description: Low level viremia is defined as a VL measurement greater than (>) 50 - <200 c/mL for pre-treated participants. For naive participants, a VL measurement between >50 to <200 c/mL after initial suppression of <50 c/mL was evaluated.
Time Frame: At Month 6 and years 1, 2 and 3
Population: The analysis was performed on the ES, which includes all participants from the FAS except those excluded for various reasons, such as protocol violations and participant withdrawal. As per protocol, data for this outcome measure were analyzed separately for ART-naive and Pre-treated participants, as the variable required different and/or additional response options depending on prior treatment status.
Measure: Number; unit: Percentage of participants
Groups:
- ART-naive Participants: Antiretroviral treatment (ART) naïve HIV-1 positive participants for whom DTG+3TC is indicated according to local label.
- Pre-treated Participants: Pre-treated HIV-1 positive participants for whom DTG+3TC is indicated according to local label.
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants
  Month 6 | 3.2 | 1.8
  Year 1 | 3.2 | 1.5
  Year 2 | 6.5 | 0.9
  Year 3 | 3.2 | 1.8

2. Secondary Outcome: Percentage of Participants With Virologic Rebound
Description: Virologic rebound is defined as 2 consecutive VL measurements >=200 c/mL after suppression. Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants | 3.4 | 0.3

3. Secondary Outcome: Percentage of Participants With Treatment Switch Due to Virologic Reasons or Due to Intolerability
Description: The intolerability was determined at the discretion of the physician. Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants
  Virologic reasons | 3.2 | 1.5
  Intolerability | 9.7 | 3.6

4. Secondary Outcome: Percentage of Participants With Missed Monthly Doses
Description: Participants were prompted to give an estimate of their level of adherence in a single-item question part of their self-assessment questionnaires. 0-2 missed doses, 3-4 missed doses, 5-6 missed doses, and >6 missed doses were reported.
Time Frame: At years 1, 2 and 3
Population: The analysis was performed on the ES, which includes all participants from the FAS except those excluded for various reasons, such as protocol violations and participant withdrawal.
Measure: Number; unit: Percentage of participants
Arm/Group | Total Participants
Number analyzed (Participants) | 228
Percentage of participants
  At Year 1 - 0-2 missed doses: number analyzed (Participants) | 185
  At Year 1 - 0-2 missed doses | 93
  At Year 1 - 3-4 Missed doses | 14
  At Year 1 - 5-6 Missed doses: number analyzed (Participants) | 185
  At Year 1 - 5-6 Missed doses | 1
  At Year 1 - >6 Missed doses: number analyzed (Participants) | 185
  At Year 1 - >6 Missed doses | 1
  At Year 2 - 0-2 missed doses: number analyzed (Participants) | 208
  At Year 2 - 0-2 missed doses | 98
  At Year 2 - 3-4 Missed doses: number analyzed (Participants) | 208
  At Year 2 - 3-4 Missed doses | 1
  At Year 2 - 5-6 Missed doses: number analyzed (Participants) | 208
  At Year 2 - 5-6 Missed doses | 1
  At Year 2 - >6 Missed doses: number analyzed (Participants) | 208
  At Year 2 - >6 Missed doses | 1
  At Year 3 - 0-2 missed doses | 99
  At Year 3 - 3-4 Missed doses: number analyzed (Participants) | 185
  At Year 3 - 3-4 Missed doses | 1
  At Year 3 - 5-6 Missed doses | 0
  At Year 3 - >6 Missed doses | 0

5. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: The analysis was performed on the Safety Analysis Set, which includes all ES participants who received at least one dose, plus those excluded from ES due to withdrawal but with available safety data. As per protocol, data for this outcome measure were analyzed separately for ART-naive and Pre-treated participants, as the variable required different and/or additional response options depending on prior treatment status.
Measure: Number; unit: Count of events
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 337
Count of events | 1 | 78

6. Secondary Outcome: Frequency of Serious Adverse Events
Description: as for outcome 5
Time Frame: From Baseline until Year 3
Population: as for outcome 5
Measure: Number; unit: Events per person-years
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 337
Events per person-years | 0.01 | 0.09

7. Secondary Outcome: Number of Serious and Non-serious Adverse Drug Reactions (ADRs)
Description: An ADR is defined as a noxious and unintended response to a medicinal investigational product related to any dose where at least a reasonable possibility, i.e. the relationship cannot be ruled out. A serious ADR is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 5
Measure: Number; unit: Count of events
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 337
Count of events
  Serious ADRs | 5 | 27
  Non-serious ADRs | 5 | 22

8. Secondary Outcome: Frequency of Any Adverse Drug Reactions
Description: Any = serious and non-serious ADRs. An ADR is defined as a noxious and unintended response to a medicinal investigational product related to any dose where at least a reasonable possibility, i.e. the relationship cannot be ruled out. A serious ADR is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 5
Measure: Number; unit: events per person-years
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 337
events per person-years | 0.06 | 0.03

9. Secondary Outcome: Discontinuation Rates Due to Adverse Drug Reactions
Description: Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: The analysis was performed on the Safety Analysis Set, which includes all ES participants who received at least one dose, plus those excluded from ES due to withdrawal but with available safety data.
Measure: Number; unit: Percentage of participants
Arm/Group | Total Participants
Number analyzed (Participants) | 368
Percentage of participants | 3.9

10. Secondary Outcome: Percentage of Participants With VL > 50 c/mL With Emergent Resistance Mutations
Description: Newly identified resistance-associated mutations, including those detected before initiating treatment with DTG+3TC and most recent HIV-RNA levels.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants | 0 | 0.3

11. Secondary Outcome: Change in Lipid Laboratory Values
Description: The following lipid parameters are presented: total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: At years 1, 2 and 3 compared to Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
mg/dL
  At Year 1 - Total cholesterol | 13.0 [-2.0 to 24.0] | -4.0 [-21.0 to 15.0]
  At Year 2 - Total cholesterol | -1.0 [-12.0 to 43.0] | -1.0 [-22.0 to 14.0]
  At Year 3 - Total cholesterol | 8.5 [-9.0 to 14.0] | -6.0 [-39.0 to 14.0]
  At Year 1 - LDL cholesterol | 3.5 [-10.0 to 17.0] | 0.0 [-16.0 to 16.0]
  At Year 2 - LDL cholesterol | 2.0 [-7.0 to 27.0] | 2.0 [-18.0 to 20.0]
  At Year 3 - LDL cholesterol | 8.5 [-16.5 to 19.5] | 0.0 [-28.0 to 17.4]
  At Year 1 - HDL cholesterol | 1.0 [-3.0 to 5.0] | 0.0 [-5.0 to 4.0]
  At Year 2 - HDL cholesterol | 3.0 [-2.0 to 5.0] | 0.0 [-4.0 to 5.0]
  At Year 3 - HDL cholesterol | 3.0 [-4.0 to 8.0] | -1.0 [-6.0 to 4.0]
  At Year 1 - Triglycerides | 6.0 [-12.0 to 39.0] | -3.0 [-43.0 to 34.5]
  At Year 2 - Triglycerides | 14.0 [-18.0 to 27.0] | -6.5 [-51.0 to 33.0]
  At Year 3 - Triglycerides | -16.5 [-69.0 to 47.0] | -13.0 [-47.0 to 29.0]

12. Secondary Outcome: Percentage of Participants With Reasons for Therapy Switch to DTG+3TC
Description: The primary reasons for therapy switch are side effects of previous ART, low potential for interaction, preference of a 2-drug regime, tolerability profile of DTG+3TC, pill size, easy to take (once daily, independent of meals), patient's preference, and other.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: At Baseline
Population: The analysis was performed on the ES, which includes all participants from the FAS except those excluded for various reasons, such as protocol violations and participant withdrawal. Only Pre-treated participants were included, as the instrument presents the reasons for therapy switch, which requires a previous regimen before DTG + 3TC.
Measure: Number; unit: Percentage of participants
Arm/Group | Pre-treated Participants
Number analyzed (Participants) | 335
Percentage of participants
  Side effects of previous ART | 39
  Low potential for interaction | 14
  Preference of a 2-drug regime | 62
  Tolerability profile of DTG+/3TC | 26
  Pill size | 1
  Easy to take (once daily, independent of meals) | 21
  Patient's preference | 21
  Other | 15

13. Secondary Outcome: Percentage of Participants With Reasons for DTG+3TC Therapy Initiation
Description: The primary reasons for therapy switch are low potential for interaction, preference of a 2-drug regime, prevention of potential long-term toxicities of other therapies, tolerability profile of DTG+3TC, easy to take (once daily, independent of meals), and other.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: At Baseline
Population: The analysis was performed on the ES, which includes all participants from the FAS except those excluded for various reasons, such as protocol violations and participant withdrawal. Only ART-naive participants were included, as the instrument presents the reasons for therapy initiation, which requires no previous regimen before DTG + 3TC.
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants
Number analyzed (Participants) | 31
Percentage of participants
  Low potential for interaction | 3
  Preference of a 2-drug regime | 45
  Prevention of potential long-term toxicities of other therapies | 6
  Tolerability profile of DTG+/3TC | 6
  Easy to take (once daily, independent of meals) | 16
  Other | 23

14. Secondary Outcome: Change in Treatment Satisfaction
Description: The change in treatment satisfaction is based on the HIV Treatment Satisfaction questionnaire (HIV TSQ). The HIV TSQ is a 10-item-self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience and flexibility. In treatment satisfaction score ranges from 0-60, where higher the score, greater the satisfaction with treatment. Individual item scores which included All rate score ranging from 0 (very dissatisfied, inconvenient, inflexible) to 6 (very satisfied, convenient, flexible), in case of general satisfaction, there will be 10 items which will be summed to produce a score ranging from 0 to 30, with higher the score greater the satisfaction with subscale. For lifestyle scale with 8 items which will be summed to produce a score ranging from 0 to 30, with higher the score greater the satisfaction with subscale.
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: At years 1, 2 and 3 compared to Baseline
Population: The analysis was performed on the ES, including all FAS participants except those excluded for reasons such as protocol violations or withdrawal. Only Pre-treated participants were included, as the instrument compares to prior treatment, which requires a previous regimen before DTG + 3TC. Only those who completed the HIV TSQ at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pre-treated Participants
Number analyzed (Participants) | 220
Scores on a scale
  At Year 1 | 1.0 [0.0 to 6.0]
  At Year 2: number analyzed (Participants) | 179
  At Year 2 | 1.0 [0.0 to 5.0]
  At Year 3: number analyzed (Participants) | 169
  At Year 3 | 1.0 [-1.0 to 5.0]

15. Secondary Outcome: Change in Symptom Distress
Description: The change in symptom distress is based on the HIV Symptom Distress Module (SDM) questionnaire. The SDM is a 20-item self-reported tool that assesses the presence and distress of symptoms related to HIV or its treatment. It includes sub-scales for treatment satisfaction and individual satisfaction with treatment changes. The treatment satisfaction score sums all items, ranging from +30 (greater improvement) to -30 (greater deterioration). Individual item scores range from +3 (much more satisfied, convenient, flexible) to -3 (much less satisfied, convenient, flexible). General satisfaction and lifestyle scores sum all items, ranging from +15 (greater improvement) to -15 (greater deterioration).
  Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: At years 1, 2 and 3 compared to Baseline
Population: The analysis was performed on the ES, which includes all participants from the FAS except those excluded for various reasons, such as protocol violations or withdrawal. As per protocol, data for this outcome measure were analyzed separately for ART-naive and Pre-treated participants, as the variable required different and/or additional response options depending on prior treatment status. Only participants who completed the HIV SDM questionnaire at the specified time points, were analyzed.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 6 | 128
Scores on a scale
  At Year 1 | -2.0 [-9.0 to 2.0] | -2.0 [-7.0 to 2.0]
  At Year 2: number analyzed (Participants) | 5 | 110
  At Year 2 | 3.0 [-3.0 to 6.0] | 0.0 [-6.0 to 5.0]
  At Year 3: number analyzed (Participants) | 6 | 94
  At Year 3 | -1.0 [-6.0 to 1.0] | 0.0 [-5.0 to 5.0]

16. Secondary Outcome: Number of HIV-RNA Monitoring Measures
Description: Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: measurements/year
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
measurements/year | 4 [3.5 to 4.2] | 4 [3.5 to 4.2]

17. Secondary Outcome: Percentage of Participants Referred to Another Medical Specialist
Description: Baseline represents the last visit before the start of therapy with DTG+3TC.
Time Frame: From Baseline until Year 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants | 38.7 | 71.6

18. Primary Outcome: Percentage of Participants With Sustained Virologic Suppression
Description: Virologic suppression is defined as a viral load (VL) less than (<) 50 copies (c)/mL or, if between 50-200 c/mL, with a subsequent next available measurement <50 c/mL (within 120 days).
Time Frame: At Year 3
Population: The analysis was performed on the Effectiveness Set (ES) which includes all participants from the Full Analysis Set (FAS) except those excluded for various reasons, such as protocol violations and participant withdrawal. As per protocol, data for this outcome measure were analyzed separately for ART-naive and Pre-treated participants, as the variable required different and/or additional response options depending on prior treatment status.
Measure: Number; unit: Percentage of participants
Arm/Group | ART-naive Participants | Pre-treated Participants
Number analyzed (Participants) | 31 | 335
Percentage of participants
  HIV-RNA <50 c/mL | 67.7 | 75.5
  HIV-RNA 50-200 c/mL & subsequent measurement <50 c/mL | 0 | 0.3

ADVERSE EVENTS:
Time Frame: Serious adverse events and all-cause mortality were collected from Baseline until Year 3. Baseline representing the last visit before the start of therapy with DTG+/3TC.
Description: In line with the pharmacovigilance plan and SOP for safety data collection in post-marketing non-interventional studies not classified as PASS, only serious and/or drug-related adverse events were required to be collected. Therefore, other adverse events were not collected for this study.
  The analysis was performed on the Safety Analysis Set. As per protocol, SAEs and all-cause mortality data were analyzed separately for ART-naive and pre-treated participants.
Arm/Group | ART-naive Participants | Pre-treated Participants
All-Cause Mortality (participants affected / at risk) | 0/31 | 2/337
Serious Adverse Events (participants affected / at risk) | 1/31 | 78/337
Other Adverse Events (participants affected / at risk) | 0/31 | 0/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ART-naive Participants (N=31) | Pre-treated Participants (N=337)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Fanconi syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Family stress (Social circumstances) | 0 (0) | 1 (1)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03754803/Prot_SAP_000.pdf